CLINICAL TRIAL: NCT04228406
Title: Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Efficacy Evaluation of the Selective c-MET Inhibitor GST-HG161 in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Efficacy Evaluation of GST-HG161
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cosunter Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GST-HG161-I
Record Dates: First submitted 2020-01-07; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Solid Tumor; C-Met Mutation-Related Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GST-HG161 (Experimental): There are 7 dose cohorts, including60mg, 150mg, 300mg, 450mg, 600mg, 750mg, 900mg QD in the dose escalation stage and GST-HG161 will be administered orally to patients once daily for each dose cohort. Recommended dose in the dose expansion stage will be determined by the results in the dose escalation stage .
  Interventions: Drug: GST-HG161

INTERVENTIONS:
Drug: GST-HG161 — There are 7 dose cohorts, including60mg, 150mg, 300mg, 450mg, 600mg, 750mg, 900mg QD in the dose escalation stage and GST-HG161 will be administered orally to patients once daily for each dose cohort. Recommended dose in the dose expansion stage will be determined by the results in the dose escalation stage .
  Other Names: selected C-MET Inhibitor

SUMMARY:
Safety, tolerability, pharmacokinetic characteristics, and preliminary efficacy evaluation of the selective c-MET inhibitor GST-HG161 in patients with advanced or metastatic solid tumors: An open, single and multiple administration, dose escalation, and expanded phase I trial

DETAILED DESCRIPTION:
This is a phase I trial to evaluate safety, tolerability, pharmacokinetic characteristics, and preliminary efficacy GST-HG161.

There are 7 dose cohorts, including60mg, 150mg, 300mg, 450mg, 600mg, 750mg, 900mg QD in the dose escalation stage and GST-HG161 will be administered orally to patients once daily for each dose cohort. Recommended protocal in the dose expansion stage will be determined by the results in the dose escalation stage .

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study and sign the informed consent;
2. Aged >=18 years;
3. Patients with advanced or metastatic solid tumors diagnosed histologically or cytologically, and no approved standard treatment regimen or no efficacy or intolerance to standard treatment regimen;
4. Patients with solid tumors confirmed c-Met positive by testing. The definition of c-Met positive is: 1) IHC expression of c-Met (positive criteria : 1+ and above); 2) FISH amplification of c-Met (positive criteria: Ratio>=1.8), any positive of the above two methods can be enrolled into the group;
5. The investigators evaluate according to RECIST v1.1, subjects must have at least one evaluable focus;
6. Performance status 0 or 1 based on ECOG scale;
7. Adequate bone marrow and major organ functions:

   Bone marrow: Hemoglobin>=9.0 g/dL, absolute count of neutrophils>1.5x10^9/L, platelet≥75x10^9/L; Coagulation function: Prothrombin time (PT)<=1.5 ULN, international normalized ratio (INR)<=1.5 ULN; Hepatic function: Total bilirubin<=1.5 ULN, ALT<=2.5 ULN, AST<=2.5 ULN; For patients with hepatic metastases or hepatoma, total bilirubin<=2 ULN, ALT<=5 ULN, AST<=5 ULN are allowed; Renal function: Serum creatinine<1.5 ULN, creatinine clearance rate>50mL/min; Other laboratory inspection indexes: Lipase 1.5 ULN, amylase<1.5 ULN, albumin>=28g/L;
8. Expected survival time>=12 weeks;
9. Fertile men and women must agree to carry out birth control with effective methods for a period of 180 days from the signing of the informed consent form until the last administration of investigational drug. Fertile women include premenopausal women and women 2 years before menopause. Fertile women must have a negative pregnancy test within 7 days (including) before the first dose of the investigational drug;
10. Subjects or their legal representatives are able to communicate well with the investigators and complete the study in accordance with protocol.

Exclusion Criteria:

1. Patients with clinical symptoms of brain metastasis, spinal cord compression, carcinomatous meningitis, or other evidence showing that the brain or spinal cord metastasis has not been controlled, and patients not suitable for the group judged by the investigators;
2. Obvious basic cardiovascular diseases, including the following conditions: Prolonged QT/QTcF interval in baseline ECG (QTcF >480ms); Severe abnormalities in baseline ECG, including rhythm, conduction, and form. For example, complete left bundle branch block, degree III atrioventricular block, etc.; Cardiovascular abnormalities identified within 6 months, such as myocardial infraction, arrhythmia, angina, angioplasty, stent implantation, coronary artery bridging, congestive heart failure, etc.; Left ventricular ejection fraction is lower than the minimum normal value showed by cardiac ultrasound; Uncontrolled hypotension or uncontrolled hypertension;
3. Digestive tract disorder that affect clinical trials, such as: Intractable hiccups, nausea, emesis, etc.; Chronic digestive diseases: Crohn's disease, ulcerative colitis, etc.; Dysphagia;
4. Patients with a history of other serious underlying diseases, such as: A definite history of neurological or psychiatric disorders, including epilepsy or dementia; Patients with active hepatitis B (HBV-DNA>1000 copy number/mL), or hepatitis C virus antibody or HCV-RNA positive, or infected with human immunodeficiency virus (HIV); A history of organ transplantation; Severe infection;
5. Pregnant or lactating women;
6. Received chemotherapy, radiation therapy, hormonal therapy, biological therapy or other anti-tumor treatment within 4 weeks (from the last medication of mitomycin and nitrosoureas for at least 6 weeks, from the last medication of fluorouracil oral drugs, such as Tegafur, Capecitabine for at least 2 weeks), or the treatment is still within 5 half-life period;
7. The adverse reactions of previous anti-tumor treatments have not recovered to CTCAE 5.0 level<=1 (except for hair loss);
8. Participated in other clinical trials as a subject within 4 weeks prior to this study;
9. The investigators determine ineligible to participate in the clinical trial for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
DLT (Dose-Limiting Toxicity) | Up to 27 days
  DLT was defined as one of the following adverse events (AEs) observed in 27 days: Grade 4 hematologic AE; Grade >=3 febrile neutropenia; Grade 3 thrombocytopenia with bleeding; Grade >=3 nausea, emesis, diarrhea and constipation, despite optimal treatment; Grade >=3 non-hematological AE.
MTD (Maximum Tolerated Dose) | Up to 27 days
  MTD was defined as the dose level at which 1 out of 6 subjects or no one experienced a DLT.

SECONDARY OUTCOMES:
Area Under Curve (AUC) | Measured on 0,1, 2, 4, 6, 8, 12, 24 and 48 hours in single-dosing stage and pre-administration of day 6, day 13, day 20 and 0, 2, 4, 6, 8,12 and 24 hours of Day27 in the multiple-dosing stage.
  Plasma samples were collected at different points for pharmacokinetic analysis
Peak Plasma Concentration (Cmax) | Measured on 0,1, 2, 4, 6, 8, 12, 24 and 48 hours in single-dosing stage and pre-administration of day 6, day 13, day 20 and 0, 2, 4, 6, 8,12 and 24 hours of Day27 in the multiple-dosing stage.
  Plasma samples were collected at different points for pharmacokinetic analysis
Cl/F | Measured on 0,1, 2, 4, 6, 8, 12, 24 and 48 hours in single-dosing stage and pre-administration of day 6, day 13, day 20 and 0, 2, 4, 6, 8,12 and 24 hours of Day27 in the multiple-dosing stage.
  Plasma samples were collected at different points for pharmacokinetic analysis
T1/2 | Measured on 0,1, 2, 4, 6, 8, 12, 24 and 48 hours in single-dosing stage and pre-administration of day 6, day 13, day 20 and 0, 2, 4, 6, 8,12 and 24 hours of Day27 in the multiple-dosing stage.
  Plasma samples were collected at different points for pharmacokinetic analysis
ORR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 months
  Objective response rate (ORR) is defined as the proportion of subjects with complete or partial response as determined by the investigator using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 months
  PFS(Progression-Free-Survival) was the time from randomization until the date of objectively determined progressive disease (PD) or death due to any cause, whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: JI LI, PHD, Principal Investigator — Shanghai Oriental Hospital ,China
Locations (1):
- Shanghai Oriental Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No